CLINICAL TRIAL: NCT06146075
Title: Assessing Engagement Patterns and Participation Trends in Individuals Joining Anorexia Clinical Trials
Brief Title: Insights Into Participating in Clinical Studies for Anorexia
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 65794646
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Anorexia
Keywords: anorexia
MeSH Terms: conditions — Anorexia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials centered on anorexia serve a pivotal function in assessing the safety and effectiveness of emerging treatments for this condition.

The primary aim revolves around meticulously scrutinizing both trial completion rates and instances of voluntary withdrawal within specific patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years old and ability to provide written informed consent obtained prior to participation in the study and any related procedures being performed
* Diagnosis of anorexia
* No prior treatment for anorexia

Exclusion Criteria:

* Pregnant or lactating women
* Any serious and/or unstable pre-existing medical disorders
* Patients receiving any other investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anorexia patients who are actively considering enrolling in a clinical trial for the said condition, but have not yet completed enrollment and randomization phases.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients who decide to enroll in an anorexia clinical research | 3 months
Rate of patients who remain in an anorexia clinical trial to trial completion | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Michael, Study Director — Power Life Sciences Inc.
Locations (1):
- Power Life Sciences, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Peters K, Meule A, Voderholzer U, Rauh E. Effects of interval-based inpatient treatment for anorexia nervosa: An observational study. Brain Behav. 2021 Nov;11(11):e2362. doi: 10.1002/brb3.2362. Epub 2021 Sep 20. PMID 34543514
- [Background] Matsuo N, Morita T, Matsuda Y, Okamoto K, Matsumoto Y, Kaneishi K, Odagiri T, Sakurai H, Katayama H, Mori I, Yamada H, Watanabe H, Yokoyama T, Yamaguchi T, Nishi T, Shirado A, Hiramoto S, Watanabe T, Kohara H, Shimoyama S, Aruga E, Baba M, Sumita K, Iwase S. Predictors of responses to corticosteroids for anorexia in advanced cancer patients: a multicenter prospective observational study. Support Care Cancer. 2017 Jan;25(1):41-50. doi: 10.1007/s00520-016-3383-z. Epub 2016 Aug 18. PMID 27539132
- [Background] Tanahashi T, Kawai K, Tatsushima K, Saeki C, Wakabayashi K, Tamura N, Ando T, Ishikawa T. Purging behaviors relate to impaired subjective sleep quality in female patients with anorexia nervosa: a prospective observational study. Biopsychosoc Med. 2017 Aug 16;11:22. doi: 10.1186/s13030-017-0107-7. eCollection 2017. PMID 28824707

DOCUMENTS (1):
  • Informed Consent Form (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/75/NCT06146075/ICF_000.pdf